CLINICAL TRIAL: NCT02827162
Title: Association of Host Genetics With Vaccine Efficacy, and Evaluation of Immune Correlates of Risk From the First Proof of Concept Efficacy Study With a Tetravalent Dengue Vaccine
Brief Title: Association of Host Genetics With Vaccine Efficacy and Study of Immune Correlates of Risk From a Tetravalent Dengue Vaccine
Status: Completed | Type: Observational
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: CYD59; U1111-1127-7875 (Other: WHO)
Record Dates: First submitted 2016-06-29; First posted 2016-07-11 (Estimated); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Dengue Fever; Dengue Haemorrhagic Fever
Keywords: Dengue Fever; Dengue Haemorrhagic Fever; Tetravalent Dengue Vaccine
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Case D1: Subject having experienced a Virologically confirmed dengue infection, from the first injection until the end of the active phase, excluding Case D3 subjects
- Case D3: Subject having experienced a Virologically confirmed dengue infection, from 28 days after the third injection until the end of the Active Phase of the proof of concept (PoC) efficacy study
- Control I: Subject having not experienced a Virologically confirmed dengue infection in the Active Phase of the PoC efficacy study, and belonging to the PoC efficacy study immunogenicity subset
- Control E: Subject having not experienced a Virologically confirmed dengue infection in the Active Phase of the PoC efficacy study, and not belonging to the PoC efficacy study immunogenicity subset

SUMMARY:
Primary objectives:

* To assess how dengue vaccine efficacy varies across participant subgroups regarding polymorphism in human leukocyte antigen (HLA) alleles of interest.
* To assess the association between HLA alleles and, serotype-specific neutralization antibody titers and summary neutralization measure in the vaccine and placebo groups.
* To assess the association between the polymorphism in HLA alleles of interest and susceptibility to Dengue fever and Dengue Haemorrhagic fever.

Secondary objectives:

* To assess whether dengue serotype-specific neutralizing antibody titers and associated summary neutralization measure at 28 days post-dose 3 are related to the rate of occurrence of symptomatic Virologically-confirmed dengue infection after post-dose 3
* To evaluate whether the dengue serotype-specific neutralizing antibody and associated summary neutralization measure at 28 days post-dose 3 are related to the level of vaccine efficacy against dengue viruses after post-dose 3.

DETAILED DESCRIPTION:
The enrolled population will include both, virologically-confirmed (VC) dengue cases and subjects not having experienced a VC dengue infection (control subjects) from the first Proof of Concept efficacy study conducted in Thailand Analyses for correlates will be performed on samples collected in the context of the first proof of concept efficacy study. Sequencing of dengue viruses will also be done on samples collected within the same context. Immunogenetic testing will be performed on saliva samples collected at the study enrollment visit.

No intervention or vaccine will be provided or administered as part of this study.

ELIGIBILITY:
Inclusion Criteria:

* Subject currently enrolled in, or having recently finished, CYD57 (NCT01983553; long-term safety follow-up study of the first PoC efficacy study), included in the subjects list provided by the Sponsor, with or without past experience of virologically confirmed dengue.
* For children 7 to < 18 years. Assent form (AF) has been signed and dated by the subject, and informed consent form (ICF) has been signed and dated by the parents or another legally acceptable representative and by independent witness, as per local Ethics Committee (EC) requirement. For subjects ≥ 18 years. ICF has been signed and dated by the subject and by independent witness, as per local EC requirement.
* Subject (and parent(s) / legally acceptable representative for subject < 18 years) are able to attend the scheduled visit and can comply with all study procedures.

Exclusion Criteria:

* Any illness that, in the opinion of the Investigator, might interfere with study procedures.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Participants will include both, virologically-confirmed (VC) dengue cases and subjects not having experienced a VC dengue infection (control subjects) from the first Proof of Concept efficacy study CYD57 (NCT01983553) conducted in Thailand
Sampling Method: Non-Probability Sample
Enrollment: 334 (Actual)
Dates: Start 2016-03-29 (Actual); Primary Completion 2016-04-27 (Actual); Study Completion 2016-04-27 (Actual)

PRIMARY OUTCOMES:
Number of Symptomatic Virologically confirmed dengue cases having occurred during the Active Phase of the first proof of concept efficacy study after post dose 1 | 28 days post-injection 1 up to 4 years (the end of the Active phase)
  A symptomatic Virologically confirmed (VC) dengue case is defined as (i) Acute febrile illness with fever lasting for at least 1 day (temperature ≥37.5°C measured at least twice with an interval of at least 4 hours), and (ii) VC by reverse transcriptase polymerase chain reaction (RT PCR) and / or dengue non structural protein 1 (NS1) enzyme linked immunosorbent assay (ELISA) Antigen test
Neutralizing Antibody level against each of the four parental dengue virus serotype strains of Sanofi Pasteur's dengue vaccine constructs measured at 28 days post dose 3 | 28 days post-dose 3 (1 year post-dose 1)
Number of probable Dengue fever and Dengue Hemorrhagic Fever grade I, II, III, and IV occurring during the Active Phase of the first PoC efficacy study after post dose 1. | Up to 6 months post-dose 1
  Probable Dengue fever is an acute febrile illness with two or more of the following manifestations: Headache, Retro orbital pain, Myalgia, Arthralgia, Rash, Haemorrhagic manifestations, and Leukopaenia

SECONDARY OUTCOMES:
Number of Symptomatic Virologically confirmed dengue cases having occurred during the Active Phase of the first proof of concept efficacy study after post dose 3 | 28 days post-injection 3 up to 4 years (end of the Active phase)
  A symptomatic Virologically confirmed (VC) dengue case is defined as (i) Acute febrile illness with fever lasting for at least 1 day (temperature ≥37.5°C measured at least twice with an interval of at least 4 hours), and (ii) VC by reverse transcriptase polymerase chain reaction (RT PCR) and / or dengue non structural protein 1 (NS1) enzyme linked immunosorbent assay (ELISA) Antigen test
Neutralizing Antibody level against each of the four parental dengue virus serotype strains of Sanofi Pasteur's dengue vaccine constructs measured at post dose 3 | Post-dose 3 (1 year post-dose 1)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur SA
Locations (1):
- Investigational Site, Ratchaburi, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Result] Geretz A, Ehrenberg PK, Bouckenooghe A, Fernandez Vina MA, Michael NL, Chansinghakule D, Limkittikul K, Thomas R. Full-length next-generation sequencing of HLA class I and II genes in a cohort from Thailand. Hum Immunol. 2018 Nov;79(11):773-780. doi: 10.1016/j.humimm.2018.09.005. Epub 2018 Sep 19. PMID 30243890
- [Derived] Thomas R, Chansinghakul D, Limkittikul K, Gilbert PB, Hattasingh W, Moodie Z, Shangguan S, Frago C, Dulyachai W, Li SS, Jarman RG, Geretz A, Bouckenooghe A, Sabchareon A, Juraska M, Ehrenberg P, Michael NL, Bailleux F, Bryant C, Gurunathan S. Associations of human leukocyte antigen with neutralizing antibody titers in a tetravalent dengue vaccine phase 2 efficacy trial in Thailand. Hum Immunol. 2022 Jan;83(1):53-60. doi: 10.1016/j.humimm.2021.09.006. Epub 2021 Oct 8. PMID 34635391